CLINICAL TRIAL: NCT06207136
Title: Canadian Parkinson's Microbiome Initiative: a Pilot Phase 2 Feasibility Randomized Controlled Trial of the MIND Diet in Parkinson's Disease
Brief Title: Microbiome and Diet in Parkinson's Disease
Acronym: PD-Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Weston Family Foundation (Other)
Responsible Party: Principal Investigator, Silke Cresswell, Principal Investigator, Associate Professor Medicine, MD, FRCPC, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H23-03933
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Diet, Healthy; Gut Microbiome; Gastrointestinal Microbiome
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Intervention diet versus standard diet
Who Masked: Participant, Investigator
Masking Description: Diet groups will be labelled without reference to the specific diet allocation (example: "Yellow cooking group" or "Blue cooking group") for all participant communication.
  Random assignment to either:
  1. the active intervention diet group, or
  2. the standard-of-care diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention healthy diet (Experimental): Participants in the active intervention group will have specific diet advice delivered with motivational and behaviour-change techniques and will learn relevant cooking skills in remotely-delivered group cooking classes (via Zoom).
  Interventions: Other: Mediterranean-style diet
- Standard diet (Active Comparator): The active control group will focus on an energy-adequate diet considered standard-of-care but similar to the participant's baseline diet. The control dietary intervention group will receive general diet advice and standard care and will receive instruction in cooking skills delivered in remote group cooking classes (via Zoom).
  Interventions: Other: Mediterranean-style diet

INTERVENTIONS:
Other: Mediterranean-style diet — Coaching in the intervention diet group will promote higher consumption of healthier foods and cooking oils, while discouraging processed foods.

SUMMARY:
The goal of this pilot study is to examine the feasibility and effects of an 18-month intervention diet compared to an active control diet (standard diet) in those living with Parkinson's Disease (PD), without dementia.

Research has shown that eating components of Mediterranean diets are associated with a 30% lower risk to develop PD and a 40% lower mortality rate in those living with PD. Diet may influence the gut and microbiomes, thus may affect PD risk and progression.

This study will examine how easy it will be to adhere to a certain type of diet for 18 months and what changes may occur in the gut microbiome and in PD symptoms on a specific diet during that time.

The study will involve in-person study visits at UBC as well as online diet coaching sessions and online group cooking classes over Zoom.

This is a randomized study, meaning that participants will be assigned by chance to either the Mediterranean-style diet group or the standard diet group for the duration of the 18 months.

This pilot study will also examine recruitment rates and retention, in order to prepare for a larger future study.

DETAILED DESCRIPTION:
Those meeting general eligibility criteria and are agreeable, will come to the University of British Columbia (UBC) for an onsite Screening visit to sign the consent form, review eligibility, and complete assessments. If the additional study criteria is met during the Screening and the 4-week run-in phase, an onsite Baseline assessment will occur over 2 days. At Baseline, each participant will be randomized to either (1) the "yellow cooking group", or (2) the "blue cooking group". Participants will remain in their assigned groups for the duration of the study. Participants will also be provided with a wearable wrist device to record daily physical movement and lifestyle factors during the 18 months.

Participants in both groups will receive virtual/remote coaching (nutrition training) and group cooking classes, and also complete questionnaires (at home and in-person) and collect biological samples (urine, faecal). Onsite (in-person) visits will occur at Screening, Baseline, 3 months, 6 months, 12 months, and 18 months (end); these will include questionnaires, blood sample collections, participant feedback, magnetic resonance imaging (MRI) scans (Baseline and 18 months only).

ELIGIBILITY:
Inclusion Criteria:

Eligible if the person living with Parkinson's has/is:

1. a clinical diagnosis of PD,
2. cognitively stable (no clinical dementia),
3. between 40-80 years old,
4. able to travel to UBC for 6 onsite visits over 18 months,
5. sufficient English proficiency (coaching and cooking classes are in English only),
6. on a stable dopaminergic medication for at least one month before baseline,
7. computer and internet access at home, and can be available via video link for at least 80% of the study sessions.

Exclusion Criteria:

Not eligible, if person has/is:

1. a diagnosis of atypical parkinsonism,
2. medical or psychiatric conditions that would prevent full participation in the nutrition intervention (such as food allergies), significant dysphagia, diabetes on insulin, anti-coagulation on warfarin, and inflammatory bowel disease,
3. clinical dementia,
4. unable to complete questionnaires or understand study instructions,
5. using of immunomodulatory agents,
6. used Probiotics in the last 4 weeks prior to study start,
7. used Antibiotics in the last 3 months prior to study start,
8. contraindications for MRI.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Study retention | 18 months
  The rate of study retention and recruitment, by calculating study completion rates and mean recruitments per month. The recruitment goal is 54, with an estimated drop-out rate of 25%, with the expectation of 40 completing the 18-month intervention.

SECONDARY OUTCOMES:
Dietary adherence | 18 months
  Adherence rate will be determined by the target score of 78% on the food diary for the intervention group, and target score of 57% by the standard group.
Optimization | 18 months
  Qualitative outcomes by measuring participant input and feedback on trial design and execution as well as blinding procedures and developing standard operating procedures for clinical data collection, MRI acquisition, biological sample collection, pre-processing, storage, shipping and distribution of samples, and analyzing standard meals for nutrient content.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Appel-Cresswell, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- UBC Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No